CLINICAL TRIAL: NCT06231368
Title: The Safety and Efficacy of CNCT19 for Patients With Autoimmune Hemolytic Anemia After Failure of Three or More Lines of Therapy
Brief Title: CNCT19 for Patients With Autoimmune Hemolytic Anemia After Failure ≥3 Lines of Therapy.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Juventas Cell Therapy Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024003
Record Dates: First submitted 2024-01-22; First posted 2024-01-30 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2024-11

CONDITIONS: Autoimmune Hemolytic Anemia; Autologous CD19 CAR-T; Failure of Three or More Lines of Therapy
Keywords: Autoimmune Hemolytic Anemia; CNCT19 CAR T-Cell therapy
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CNCT19 CAR T-Cell Therapy (Experimental): Participants will receive CNCT19 cell infusion after preconditioning, and they need to be closely monitored for 24 hours following CAR-T cell infusion. Participants are advised to remain in the hospital for a minimum of 14 days following cell infusion. The duration of hospitalization and observation will be determined based on the researcher's comprehensive assessment of the subject's condition.
  Interventions: Biological: CNCT19 CAR-T cell therapy

INTERVENTIONS:
Biological: CNCT19 CAR-T cell therapy — CNCT19 was a second-generation CAR T-cell with scFv derived from clone HI19α and 4-1BB/CD3-ζ costimulatory domain.

SUMMARY:
This is a Phase 1, single-arm, open-label, dose-escalation and dose-expansion study. The main purpose is to evaluate the safety and tolerability, efficacy of CNCT19 CAR T-cell therapy in patients with autoimmune hemolytic anemia after failure of three or more lines of therapy. Participants will receive CNCT19 cell infusion after preconditioning, and they will receive a 1-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subject and/or subject's legal personal representative fully understand and voluntarily sign informed consent forms
* Male or female age ≥ 12 years
* Subjects with autoimmune hemolytic anemia or Evans syndrome after Failure ≥3 lines of therapy. The Failure of ≥3 lines of therapy meets all the following conditions: Hemoglobin less than 10g/dl and symptoms of anemia; Failure of first-line corticosteroid therapy; Failure of second-line rituximab therapy; Failure of any one or more of the third-line treatments (splenectomy, cyclosporine, cyclophosphamide, azathioprine, mycophenolate mofetil, fludarabine, bortezomib, etc.)
* Female subjects of childbearing potential must have a negative Serum HCG test within 7 days before enrollment. Subjects of childbearing potential will be required to follow contraception requirements from the time of enrollment until the 1-year follow-up after cell infusion
* Laboratory tests of adequate organ function: Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3×ULN; and have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and the blood oxygen saturation in a non-oxygenated state is >93%
* ECOG performance status ≤2
* Subject with a life expectancy of more than 3 months

Exclusion Criteria:

* History of other lymphoproliferative neoplasms
* Secondary AIHA caused by drugs or infection
* Platelets in subjects with Evans syndrome<30×10^9/L
* Pregnant or breast-feeding subjects
* Treatment with any of the following within the noted period prior to study entry: a.anti-CD20 monoclonal antibodies <12 weeks, b.sutimlimab or other marketed biologics <5 half-lives; c.plasma exchange <4 weeks; d.post-splenectomy <12 weeks
* Previously received organ or stem cell transplantation
* History of new thrombosis or organ infarction in the past 6 months
* Diagnosis of the active stage of the connective tissue disease
* Had other inherited or acquired hemolytic diseases
* Have active infections, such as sepsis, bacteremia, fungemia, uncontrolled pulmonary infection and active tuberculosis, etc.
* Positive hepatitis B surface antigen (HBsAg) or hepatitis B e antigen (HBeAg); positive hepatitis B e antibody (HBe-Ab) or hepatitis B core antibody (HBc-Ab), and the HBV-DNA copy number is above the lower limit of the measurable capacity; positive hepatitis C (HCV) antibody; positive human immunodeficiency virus (HIV) antibody; positive syphilis test
* Received major surgery within 4 weeks before screening that was assessed by the researcher as unsuitable for enrollment
* Have malignant tumors within 5 years before enrollment, except tumors with negligible risk of metastasis or death and curable tumors, such as adequately treated cervical carcinoma in situ, cutaneous basal cell carcinoma, etc.
* Have any of the following cardiovascular diseases: a.Left ventricular ejection fraction (LVEF) ≤45%, b. presence of active heart disease or congestive heart failure (New York Heart Association [NYHA] Class III or IV)), c.severe arrhythmias requiring treatment (except atrial fibrillation, paroxysmal supraventricular tachycardia), d.QTcB interval ≥450ms for men and ≥470ms for women, e.have myocardial infarction, bypass surgery, or stent placement within the 6 months before the study, f.other heart diseases judged by the researcher to be unsuitable for enrollment
* Have a history of live attenuated vaccines within 6 weeks before enrollment
* Participate in other interventional clinical studies during CNCT19 CAR T-Cell therapy, and the drug has a half-life of <5. Subjects treated with active investigational drugs or intend to participate in another clinical trial or receive treatment other than that specified in the protocol throughout the study period
* Have a history of epilepsy or other active central nervous system diseases
* Have an allergy to the ingredients of the medicine used in this study
* Previously received CAR-T cell therapy
* Patients considered to be ineligible for the study by the investigator for reasons other than the above

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-02-04 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and the severity of the adverse event | Within 12 months
  Use Common Terminology Criteria for Adverse Events (CTCAE) Version 5 to assess the adverse event

SECONDARY OUTCOMES:
Percentage of patients with hematological response | Within 24 weeks
  Hematological response is mainly evaluated by hemoglobin (Hb), laboratory Indicators of hemolysis (serum bilirubin and lactate dehydrogenase) and blood transfusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Regenerative Medicine Center, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li R, Pan H, Zhang L, Ma J, Li W, Gao Z, Fang L, Tian L, Shen Y, Yang F, Zhao J, Nie N, Li J, Wang W, Pan X, Lian Y, Li X, Peng G, Li L, Yu X, Xu C, Liu Y, Kuang Z, Huang J, Zhao X, Ge M, Liu L, Chen S, Feng Y, Chang AH, Deng B, Dai M, Huang L, Lv L, Zheng Y, Luo Y, Xiong H, Shi J. CD19 CAR T-Cell Therapy for Autoimmune Hemolytic Anemia. N Engl J Med. 2026 Jan 15;394(3):253-267. doi: 10.1056/NEJMoa2509820. PMID 41534043